CLINICAL TRIAL: NCT05113329
Title: Efficacy of Infection Control Program on Reducing Tracheostomy Tube Colonization With Biofilm Producing Antimicrobial Resistant Bacteria
Brief Title: Infection Control Program in Tracheostomized Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa Aref, Principal Investigator, Assiut University
Other Study IDs: Infection prevention & control
Record Dates: First submitted 2021-10-18; First posted 2021-11-09 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Tracheostomy Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthcare-associated infections are infections that patients acquire during the course of receiving treatment for other conditions within a healthcare setting and are not present at the time of admission. Medical instrumentation increases the risk of development of HAIs. Such devices include, venous and urinary catheters, and ventilators.

Most ventilator-dependent patients undergo respiratory stabilization with an endotracheal tube in a critical care setting. Later on, translaryngeal tubes are converted to a tracheostomy to provide long-term airway access for ventilatory support.

Tracheostomy is a commonly performed airway surgery for critically ill patients. It has variable complications, a common one being secondary infection with bacteria and fungi, which in turn leads- to granulation formation in stoma and on peristomal region.

The risk factor for infection in patients with tracheostomy occurs due to exposure to large amounts of bacteria because they do not pass through the upper airway defense system.

The commonest microorganism colonizing the tracheostomy tube leading to respiratory infections include Pseudomonas aeurginosa, Acinetobacter baumanii, and methicillin resistant Staphylococcus aureus, some of these organisms are antibiotic resistant.

Biofilm formation is a unique self-protective mechanism of bacteria, protects them from host immune response and antimicrobial agents. Studies showed that more than 60% of hospital acquired infections are caused by biofilm forming bacteria on medical devices. These infections are most commonly attributed to Staphylococcus aureus, Pseudomonas, and mixed flora.

DETAILED DESCRIPTION:
Healthcare-associated infections (HAIs) are infections that patients acquire during the course of receiving treatment for other conditions within a healthcare setting and are not present or incubating at the time of admission. Medical instrumentation increases the risk of development of HAIs and most patients admitted for health care are exposed to some kind of medical device in the course of their treatment. Such devices include, but are not limited to, venous and urinary catheters, and ventilators.

Most ventilator-dependent patients first undergo respiratory stabilization with a translaryngeal endotracheal tube in a critical care setting. At some time during the course of their disease, translaryngeal tubes are converted to a tracheostomy to provide long-term airway access for ventilatory support.

Tracheostomy is a commonly performed airway surgery for critically ill patients. It is a lifesaving procedure done for mechanical ventilation, bronchopulmonary toileting and reduce pulmonary effort.

Tracheostomy tubes have a main shaft (cannula) attached to a neck plate (or flange), and cuffed tubes have a pilot balloon, which shows whether the cuff is inflated. The neck plate has a slot where ties can be placed, and fenestrated tubes can have a cuff and/or inner cannula. Their insertion is aided with an obturator.

It has variable complications, a common one being secondary infection with bacteria and fungi, which in turn leads- to granulation formation in stoma and on peristomal region. As tracheostomy tube is an indwelling prosthesis, it provides potential surface for growth of bacteria.

In tracheostomized patients, the role of the nose, nasopharynx and upper respiratory mucosa as a defensive mechanism is absent which allows bacteria to have direct access from the stoma to the respiratory tract. Infections in tracheostomy stoma, tracheobronchitis, and pneumonia are common infections that occur after tracheostomy. The risk factor for infection in patients with tracheostomy occurs due to exposure to large amounts of bacteria because they do not pass through the upper airway defense system.

There is a 20 fold increase in the development of respiratory tract infection following mechanical ventilation in tracheostomized or mechanically ventilated patients, the incidence vary between 4% and 28%. The commonest microorganism colonizing the tracheostomy tube leading to respiratory infections include Pseudomonas aeurginosa, Acinetobacter baumanii, and methicillin resistant Staphylococcus aureus, some of these organisms are antibiotic resistant which in turn increase the morbidity and costs involved.

The tracheal cannula is often be exposed to enzymes, antioxidants and bacteria found in the tracheal mucosa, thereby accelerating aggregation, increasing colonization of microorganisms and forming biofilms on the surface of the cannula. The irritation by tracheostomy tube causes local inflammatory reaction and edema leading to bacterial colonization. To avoid the lower respiratory tract infection, careful hygiene of tracheostomy is recommended. Using sterile disposable suction catheters, gentle tracheal suction, bacteria free humidifiers, less visitors are recommended. However, despite of high level of hygiene, exogenous colonization with or without subsequent infection is common.

The outer cannula of tracheostomy tubes are routinely changed for a number of reasons. Regular tube changes are thought to aid in the prevention of stoma granulation tissue formation and tube blockage but are mainly done to reduce the rates of possible infection. Biofilm formation is a commonly cited reason for regular tracheostomy tube changes despite little supporting evidence, as they have are believed to cause deterioration in the tube surfaces. Inner cannulas of tracheostomy tubes act as liners and are changed on a daily or more often basis to prevent mucous build-up. A clinical consensus statement on tracheostomy care emphasized that effective wound care for tracheostomy patients has the positive effects of reducing the infection rate, shortening the time with a tracheal tube and improving patients' life quality. Gauze or moist dressings are widely used to take care of tracheostomy wounds.

Biofilm formation is a unique self-protective mechanism of bacteria, as it protects them from host immune response and antimicrobial agents. Biofilms are complex three dimensional structures, which are composed of bacteria, living in an extracellular matrix made of polysaccharides, nucleic acids and proteins. Studies showed that more than 60% of hospital acquired infections are caused by biofilm forming bacteria on medical devices. These infections are most commonly attributed to Staphylococcus aureus, Pseudomonas, and mixed flora.

Data regarding the colonization rates of tracheostomy tubes and the antimicrobial resistance and biofilm forming potential of bacteria colonizing tracheostomy tubes in Upper Egypt is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* It includes tracheostomized adult patients (age > 16 years) from both sexes with tube in situ for more than 7 days.

Exclusion Criteria:

* Patients will be excluded if they underwent an emergency tracheostomy tube change (i.e from dislodgement or obstruction), continue to require ongoing active machine ventilation, have an active lower respiratory tract infection or are immunosuppressed

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients (age > 16 years) from both sexes with tube in situ for more than 7 days at ENT department, Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of infection control program on reducing tracheostomy tube colonization with biofilm producing antimicrobial resistant bacteria | baseline
  Assessment of infection control program performance among tracheostomized patients.
  Identify the bacteria colonizing the tracheostomy tubes and their antibiotic resistance.
  Recognize biofilm producing bacterial isolates. Characterize the exopolysaccharides encoding genes that correlate with bioflm formation.

REFERENCES:
- [Background] Mathur T, Singhal S, Khan S, Upadhyay DJ, Fatma T, Rattan A. Detection of biofilm formation among the clinical isolates of Staphylococci: an evaluation of three different screening methods. Indian J Med Microbiol. 2006 Jan;24(1):25-9. doi: 10.4103/0255-0857.19890. PMID 16505551
- [Background] Kamali E, Jamali A, Ardebili A, Ezadi F, Mohebbi A. Evaluation of antimicrobial resistance, biofilm forming potential, and the presence of biofilm-related genes among clinical isolates of Pseudomonas aeruginosa. BMC Res Notes. 2020 Jan 10;13(1):27. doi: 10.1186/s13104-020-4890-z. PMID 31924268
- [Background] Miari M, Rasheed SS, Haidar Ahmad N, Itani D, Abou Fayad A, Matar GM. Natural products and polysorbates: Potential Inhibitors of biofilm formation in Pseudomonas aeruginosa. J Infect Dev Ctries. 2020 Jun 30;14(6):580-588. doi: 10.3855/jidc.11834. PMID 32683348
- [Background] Bogiel T, Depka D, Rzepka M, Kwiecinska-Pirog J, Gospodarek-Komkowska E. Prevalence of the Genes Associated with Biofilm and Toxins Synthesis amongst the Pseudomonas aeruginosa Clinical Strains. Antibiotics (Basel). 2021 Feb 28;10(3):241. doi: 10.3390/antibiotics10030241. PMID 33670887
- [Background] Heffner JE, Hess D. Tracheostomy management in the chronically ventilated patient. Clin Chest Med. 2001 Mar;22(1):55-69. doi: 10.1016/s0272-5231(05)70025-3. PMID 11315459
- [Background] Raveendra N, Rathnakara SH, Haswani N, Subramaniam V. Bacterial Biofilms on Tracheostomy Tubes. Indian J Otolaryngol Head Neck Surg. 2022 Dec;74(Suppl 3):4995-4999. doi: 10.1007/s12070-021-02598-6. Epub 2021 May 6. PMID 33972925
- [Background] Hutauruk SM, Hermani B, Monasari P. Role of chlorhexidine on tracheostomy cannula decontamination in relation to the growth of Biofilm-Forming Bacteria Colony- a randomized controlled trial study. Ann Med Surg (Lond). 2021 Jun 10;67:102491. doi: 10.1016/j.amsu.2021.102491. eCollection 2021 Jul. PMID 34194732
- [Background] Tan CY, Chiu NC, Lee KS, Chi H, Huang FY, Huang DT, Chang L, Kung YH, Huang CY. Respiratory tract infections in children with tracheostomy. J Microbiol Immunol Infect. 2020 Apr;53(2):315-320. doi: 10.1016/j.jmii.2018.07.002. Epub 2018 Aug 9. PMID 30131258
- [Background] Kumarasinghe D, Wong EH, Duvnjak M, Smith MC, Palme CE, Riffat F. Colonization rates of tracheostomy tubes associated with the frequency of tube changes. ANZ J Surg. 2020 Nov;90(11):2310-2314. doi: 10.1111/ans.15970. Epub 2020 May 17. PMID 32419324
- [Background] Bontempo LJ, Manning SL. Tracheostomy Emergencies. Emerg Med Clin North Am. 2019 Feb;37(1):109-119. doi: 10.1016/j.emc.2018.09.010. PMID 30454773